CLINICAL TRIAL: NCT05832944
Title: Hyomental Distance Measured Ultrasonography Versus Weight-based Criteria for Laryngeal Mask Size Selection in Children. A Prospective, Randomised Controlled Study
Brief Title: Hyomental Distance Measured Ultrasonography Versus Weight-based Criteria for Laryngeal Mask Size Selection in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, AHMED ABDELAZIZ SHAMA, Assistant professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: MKSU 51-2-18
Record Dates: First submitted 2023-04-16; First posted 2023-04-27 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Laryngeal Mask Airway
Keywords: hyomental distance; children

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group HMD (30 patients) (Experimental): where the size of LMA will be according to measured hyomental distance by ultrasound as follows:
  * If Less than 2 cm: LMA size 2 will be used.
  * If 2-3 cm: LMA size 2.5 will be used.
  * If more than 3 cm: LMA size 3 will be used.
  Interventions: Device: ultrasound guided hyomental distance
- Group CONTROL (30 patients) (No Intervention): where size selection will be based on the weight guide

INTERVENTIONS:
Device: ultrasound guided hyomental distance — measuring the hyomental distance by ultrasound guidance
  Arms: Group HMD (30 patients)

SUMMARY:
* In pediatric surgery and emergencies, LMA represents a useful airway management device for routine and difficult airway management.
* Inserting an improper LMA size may result in malposition, displacement within the hypopharynx, and failed ventilation that needs repositioning.
* Selection of the size of LMA represents a major challenge for anesthesiologists, especially in children.
* The ultrasonographic measured hyomental distance showed a correlation with the length of the pharyngeal cavity.
* Optimization of the size of the inserted LMA can be confirmed either clinically, ultrasonographic or through the fiberoptic laryngoscope.
* The ultrasonographic measured hyomental distance confirmed the optimization of LMA with results comparable to that of the clinical methods and better than those of the fiberoptic laryngoscope.

DETAILED DESCRIPTION:
* The laryngeal mask airway (LMA) is classified as one of the supraglottic devices that have been extensively adopted as an adjunctive or alternative technique to tracheal intubation or mask ventilation for airway management in short-time surgery. Moreover, it is characterized by ease of placement and removal, less injury to the respiratory tract, better tolerability by patients, improved hemodynamic stability, less coughing, less sore throat, avoidance of laryngoscopy, and hands-free airway. However, it is not suitable to overcome functional airway problems and mechanical airway obstruction.
* Although the weight-based method was considered the traditional method for the selection of the optimal LMA size, a clinical practice viewed that this method is not always applicable as there is no linear correlation between the upper airway anatomy and body weight with the presence of usual individual anatomical variation.
* Fortunately, ultrasonography gave high-resolution images of the anatomic structures of the upper airway comparable to computed tomography and magnetic resonance imaging, Ultrasound measurements were applied for the hyomental distance and the hyomental distance ratio. Some studies revealed variable sensitivity and specificity.
* This prospective randomized controlled study will aim to assess the efficacy and safety of ultrasonographic measured hyomental distance in the optimization of the laryngeal mask(LMA)size selection and placement in pediatric patients Operational Design

A) Pre-anaesthetic management:

* Informed written parental consent will be taken from all participants.
* Medical history and complete clinical examination.
* Routine laboratory investigation including :

  1. CBC
  2. CRP
  3. INR, PT & PTT
* Patients will fast for at least 8 hours before surgery.
* Routine Monitoring, including heart rate (HR), oxygen saturation (SpO2) and noninvasive blood pressure (NIBP) in the pre-anaesthesia room (Base Line Data).
* A peripheral intravenous line (24-22G) will be inserted.
* A premedication of 0.01 mg/kg Atropine will be administrated IM 1 hour before surgery.

B) Induction of general anaesthesia:

* Routine monitoring, including heart rate (HR), oxygen saturation (SpO2), noninvasive blood pressure (NIBP) and continuous electrocardiography (ECG) in the operation room.
* Intravenous induction of anaesthesia will be performed using Propofol 2 mg/kg, and fentanyl 1µg/kg.
* Mechanical Ventilation: 6-8 mL/kg Tidal Volume, 10-20 bpm Respiratory Rate, end-tidal CO2 35-40 mmHg and Volume Controlled ventilation with an inspiratory-expiratory ratio of 1:2 will be initiated.
* For all patients, maintenance of anaesthesia will be performed using Sevoflurane 1-2 %. The depth of anaesthesia will be monitored according to HR.

C) Process:

1. Before starting the current study, a pilot experiment has been done, measuring the upper airway parameters of 10 children who used LMA during operation by ultrasound, investigators found that when the hyomental distance was less than 2 cm, 80% of subjects were suited for class 2 LMA and if 2-3 cm, suited for class 2.5 LMA. Additionally, size 3 LMA were fitted to the hyomental distance above 3 cm.
2. After getting ethical committee approval, and clinical trial registration, 60 pediatric participants will be scheduled for surgery using a laryngeal mask and will be divided randomly into two groups (30 in each group)

ELIGIBILITY:
Inclusion Criteria:

* Parents' acceptance
* Age: between 5-14 years
* Physical Status: American Society of Anesthesiologists (ASA) I & II)

Exclusion Criteria:

* Developmental Delay (mental and physical growth retardation).
* Hypersensitivity to any type of used drugs.
* Patient with a difficult airway ( according to thyromental height and the Mallampati test)
* Patients with a history of neck surgery
* Airway malformation.
* Upper respiratory tract infection.
* Surgeries that will take up to more than forty-five minutes.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
correct size selection of LMA | During LMA insertion (5 minutes duration)
  * A five-point scale will be used to evaluate the ease of LMA insertion from 1 to 5, considering that 1 corresponds to (inserted without resistance) and 5 corresponds to (impossible to insert).

SECONDARY OUTCOMES:
Values of oropharyngeal leak pressure (OLP) after airway management | During 30 minutes after LMA insertion
  hearing of leakage sounds from LMA
postoperative oral injury | After removal of LMA for 5 minutes
  blood adhering to the LMA surface
many insertion attempts | During LMA insertion attempts for 5 minutes
  defined as re-insertion after complete LMA removal from the oral cavity

CONTACTS AND LOCATIONS:
Overall Officials: AHMED A SHAMA, MD, Principal Investigator — Assistant professor of anesthesia in Tanta University
Locations (1):
- kafrelsheikh university, Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No